CLINICAL TRIAL: NCT04594382
Title: Monitoring Pupillary Reflex Dilatation for Optimized Postoperative Opioid Delivery Before Extubation: A Randomized Pupillometry Study
Brief Title: Monitoring Pupillary Reflex Dilatation for Optimized Postoperative Opioid Delivery Before Extubation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2063/2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Infrared Pupillometry; Postoperative Opioid Consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T30/60 (Active Comparator): Before extubation, opioid administration will be given by a single dose of opioids in case of measured PDR values of ≥12.
  Interventions: Diagnostic Test: Pupillometry-Opioid treatment
- Non-T30/60 (Active Comparator): A standardized single dose of opioid will be given intravenously before extubation, regardless of the measured pupillometry PDR values.
  Interventions: Diagnostic Test: Pupillometry -standardized opioid treatment
- Standard Care group (No Intervention): The amount of administered piritramid in the OR will be left to the discretion of the anesthesiologist attending the participant.

INTERVENTIONS:
Diagnostic Test: Pupillometry-Opioid treatment — At the end of anesthesia, before extubation, pupillometry measurements will be performed on both eyes, using the tetanus mode T30 (30mA tetanic stimulation) and T60 (60mA tetanic stimulation) and the standardized pupillary pain index (PPI) mode at the pupillometer.
  Opioid administration will be given by a single dose of piritramid (0.1 mg kg -1) in case of measured PDR values of ≥12 (high analgesic sensitivity as specified by the producer) after T30 and T60 stimulation. The pupillometry measurement will be repeated once on both eyes.
  Arms: T30/60
Diagnostic Test: Pupillometry -standardized opioid treatment — At the end of anesthesia, before extubation, pupillometry measurements will be performed on both eyes, using the tetanus mode T30 (30mA tetanic stimulation) and T60 (60mA tetanic stimulation) and the standardized pupillary pain index (PPI) mode at the pupillometer.
  A standardized single dose of piritramid (0,1 mg kg -1) will be given intravenously, regardless of the measured values. The pupillometry measurement will be repeated once on both eyes.
  Arms: Non-T30/60

SUMMARY:
The study will be designed to investigate the effect of pupillometry guided compared to non-PPI-guided postoperative pain therapy, conducted immediately at the end of surgery before extubation, on total postoperative opioid consumption during the first 2 postoperative hours after elective ear nose throat (ENT) surgery.

DETAILED DESCRIPTION:
Pupillometric pain measurements helps clinicians determine and administer the optimized amount of opioids and so avoids opioid-induced side effects.The study will be designed to investigate the effect of pupillometry guided compared to non-PPI-guided postoperative pain therapy, conducted before extubation, on total postoperative opioid consumption during the first 2 postoperative hours after elective ENT surgery.

Background The evaluation of pain intensity during the immediate postoperative period in the operating room (OR) is a key factor for post interventional pain treatment. However, this evaluation may be difficult when patients are still intubated, restricted in consciousness or are showing verbal impairment due to ENT surgery. Verbally impaired patients are at increased risk of under treatment for pain.

With rising opioid consumption, the risk of postoperative side effects like nausea and vomiting, sedation with a longer recovery time or respiratory depression increases. Especially in the cohort of ENT surgery patients, where a difficult airway is regularly presented, such side effects should be avoided. A means of predicting immediate postoperative pain after surgery and the response to opiate analgesics would therefore be highly desirable.

The pupillary dilatation reflex (PDR), measured by pupillometry, has been successfully used to assess intraoperative analgesic component of anesthetic regimes and correlates with pain intensity measured on a numeric rating scale (NRS).

Aims

Primary aim of this study is to investigate if a pupillometry-guided opioid administration immediately postoperative in the OR leads to less opioid requirement during the first 2 postoperative hours compared to a non-pupillometry-guided treatment.

Secondary aim is to evaluate postoperative pain intensity during the first 2 postoperative hours in patients after pupillometry-guided versus non-pupillometry -guided opioid therapy in the OR.

Hypotheses

The investigators hypothesis that through a targeted pain therapy based on the measurement of immediate postoperative pupillometry scores, opioid consumption and pain intensity can be reduced during the first 2 postoperative hours.

Methods

The study will be done by observing postoperative pain intensity using pupillometry in patients scheduled for elective ENT surgery, carrying out pain intervention (opioid therapy) and re-observing to verify the effectiveness of the targeted postoperative opioid administration in the OR. Pain on an 11-point verbal Likert response score and total opioid consumption will be recorded by a blinded investigator at 30-minute intervals for the initial 2 postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I-II
* able to read and understand the information sheet and to sign the consent form
* being scheduled for elective ENT surgery under general anesthesia
* age≥18 years

Exclusion Criteria:

* ASA physical status of III and above
* previous history of either drug or alcohol abuse
* difficulty to understand pain scoring system
* chronic users of analgesics or had used opioids within 12 h before surgery
* drug or alcohol abuse
* contraindications for metamizole
* preoperative topical eye medication (atropine, phenylephrine), preoperative pupil abnormality
* concomitant treatment with beta-antagonists, metoclopramide or droperidol
* implanted electronic medical devices
* dysfunction of the autonomic nervous system in relation to advanced diabetes mellitus
* ophthalmologic diseases, known pupil reflex disorders, cranial nerve lesions
* rapid sequence induction (RSI)
* neurological, psychiatric or mental disorders
* surgical procedure warranting elective postoperative ventilation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | first 2 postoperative hours
  cumulative opioid consumption within first 2 postoperative hours

SECONDARY OUTCOMES:
postoperative pain intensity | first 2 postoperative hours
  Pain on an 11-point verbal Likert response score (VAS score) recorded by a blinded investigator at 30-minute intervals for the initial 2 postoperative hours. The 11-point numeric scale ranges between 0, meaning no pain, and 10, meaning worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No